CLINICAL TRIAL: NCT06852326
Title: Designing a Tailored Primary Care Intervention to Manage the Burden of Caring for Patients Living with Alzheimer's Disease (or a Related Dementia)
Acronym: ISAMA-PP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR240112 - ISAMA-PP
Record Dates: First submitted 2025-01-31; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Primary Care; Alzheimer Disease
Keywords: care; caregiver
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group caregiver: Qualitative interviews and focus groups
- Group health professional: Qualitative interviews and focus groups
- Group academic expert: Qualitative interviews and focus groups

SUMMARY:
The design of the intervention is an ongoing process which will consist of two phases: a determination of the intervention using the Delphi-modified consensus method and an assessment of its acceptability, as described in the methodological recommendations of the Medical Research Council Guidance.

DETAILED DESCRIPTION:
First phase : determination of the intervention.

A list of proposed interventions drawn from the literature and the exploratory work will be proposed to panels of participants using the DELPHI-modified method : Rounds made up of a panel of carers, a panel of healthcare professionals in the field, and a panel of academic experts who have knowledge of the scientific literature on the subject as well as having clinical experience.

The method consists of proposing different intervention proposals and having them validated/modified using a Likert scale by scoring during different e-Delphi rounds (a paper version of the questionnaire will also be available). Following each Delphi round, a meeting will be organised with all the members of each panel to discuss the comments made during these rounds.

* Each item will be graded from 1 to 9 by each participant.
* Topics with a 70% score ≥ 7 are retained.
* Topics with a score of 70% ≤ 3 are eliminated.
* Topics scoring 70% between 4 and 6 are reformulated by the members of the scientific committee and reproposed in the following round.

It usually takes between 3-4 rounds to eliminate/validate themes.

Second phase : assessment of the acceptability of the conceived intervention.

Following this consensus, a complex intervention with several components will be determined and proposed by the scientific committee to the 3 participating CPTS (territorial professional health communities): the Asclepios and Est Cher CPTS (which had already participated in the previous exploratory studies) and the Iroise CPTS (naïve to any preliminary assessment of its needs in its territory). Quantitative data on the acceptability of the intervention will then be collected, namely :

* the number of carers who were offered or not offered the intervention
* the number of carers who benefited from the intervention in its entirety or by component
* the number of carers who refused or abandoned the intervention. Qualitative data on acceptability will also be collected through observations of voluntary carers and healthcare professionals and through interviews. Throughout the process of creating the intervention (from the Delphi rounds to the proposal of the intervention to the 3 participating CPTS), an exploration of the co-construction process and the acceptability of the intervention will be carried out using qualitative Focus Group (FG) interviews with each group involved (carers, healthcare professionals, university experts), then with each CPTS (carers and healthcare professionals from each CPTS). Depending on the results of this exploration, the intervention may be adapted by the scientific committee. This is a continuous process of evaluating the intervention, as recommended in the development of complex interventions.

The whole complex intervention thus determined will be reported using the TIDieR checklist model

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals who are members of the 3 CPTSs included and who agree to participate
* Adult informal carers of patients living with Alzheimer's disease or a related dementia from the 3 CPTS who agree to participate
* University experts: general practitioners, geriatric mobile team doctor, advanced practice nurse, clinical psychologist, biostatistical methodologist. Some of them had already taken part in the steering committee for ISAMA's exploratory qualitative and quantitative studies.

Exclusion Criteria:

- Professional carers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Determining the intervention using the DELPHI-modified method, the 30 participants will be academic experts (10 people) and people from the 2 professional communities (CPTS) that took part in the exploratory studies, Asclepios and Est Cher (10 primary healthcare professionals and 10 carers). The 10 carers will have different characteristics depending on the level of dependency and the extent of the behavioural problems of the patient they are helping, and on their family status (parent, child or other). They will also come from the care areas of the 2 CPTS, Asclepios and Est Cher.
  Concerning the qualitative sociological exploration of the process of acceptability and co-construction of the intervention, the 30 participants will be academic experts (the 10 people identified above) and people from the 3 CPTS, Asclepios, Est Cher and Iroise who tested the conceived intervention (10 healthcare professionals and 10 carers).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
description of the tailored primary care intervention to manage the burden of caring for patients living with Alzheimer's disease (or related dementia) | 12 months
  A list of interventions will be submitted to 3 panels of participants using the DELPHI method (panel of carers, panel of healthcare professionals and panel of academic experts). Each participant will rate his or her agreement with each of the proposals with a score ranging from 1 (strongly disagree) to 9 (strongly agree).
  For each proposal, the proportion of scores >= 7, the proportion of scores between 4 and 6 and the proportion of scores <=3 will be estimated. Proposals with at least 70% of ratings >= 7 are retained. Proposals with at least 70% of scores <= 3 are eliminated. Proposal with at least 70% of scores between 4 and 6 will be reformulated by the members of the scientific committee and reproposed in the following round.
  It usually takes between 3-4 rounds to eliminate/validate proposals: the complex intervention will be built on the consensus reached in theses rounds and reported using the TIDieR checklist model.

SECONDARY OUTCOMES:
acceptability of the complex intervention by carers and healthcare professionals | 6 months
  For the 3 CPTS (territorial professional health communities) participating in the study, these outcomes will be calculated:
  Number of carers to whom the intervention was offered or not Number of carers who benefited from the intervention as a whole or by component Number of carers who refused or abandoned the intervention. Qualitative data on acceptability (verbatims comments and more) will also be collected through observations and interviews of voluntary carers and healthcare professionals.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CPTS Asclepios, Amboise
  - CPTS Pays d'Iroise, Saint-Renan
  - CPTS Est Cher, Sancergues

IPD SHARING:
Plan to Share IPD: Undecided